CLINICAL TRIAL: NCT07334821
Title: Comparison of the Effectiveness of PIC Cystogram and VCUG in the Diagnosis of Vesicoureteral Reflux in Children
Brief Title: Diagnostic Performance of PIC Cystogram vs VCUG in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarik Emre Sener (Other)
Responsible Party: Sponsor-Investigator, Tarik Emre Sener, Associated Professor, Marmara University
Organization: Marmara University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MAR.UAD.0028
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Urology
Keywords: PIC Cystogram; VCUG; Vesicoureteral Reflux; Children
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single-blind (physician blinded to VCUG results)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIC cystography (Experimental)
  Interventions: Diagnostic Test: PIC cystography; Diagnostic Test: VCUG
- VCUG Group (Other)
  Interventions: Diagnostic Test: VCUG

INTERVENTIONS:
Diagnostic Test: PIC cystography — PIC cystography is performed intraoperatively during endoscopic surgery. A pediatric cystoscope is positioned adjacent to each ureteral orifice, and contrast medium is instilled by gravity from a height of 1 meter under fluoroscopic guidance. The presence and grade of vesicoureteral reflux are recorded for each renal unit. The procedure is carried out in a standardized manner by an investigator blinded to prior VCUG findings
  Arms: PIC cystography
Diagnostic Test: VCUG — VCUG performed

SUMMARY:
The goal of this interventional diagnostic clinical trial is to evaluate and compare the diagnostic effectiveness of PIC cystography and voiding cystourethrography (VCUG) for the detection of vesicoureteral reflux (VUR) in children undergoing endoscopic procedures, including those who previously underwent VCUG for urinary tract infection (UTI) or other indications, as well as children who did not require VCUG.

The main questions it aims to answer are:

Does PIC cystography detect VUR at a rate comparable to VCUG?

How well do PIC cystography and VCUG correlate in identifying low-grade versus high-grade VUR?

Researchers will compare PIC cystography findings with prior VCUG results to determine agreement between the two diagnostic methods and their ability to detect clinically relevant reflux.

Participants will:

Undergo PIC cystography performed during endoscopic surgery

Have contrast instilled near each ureteral orifice under fluoroscopic monitoring

Be evaluated for the presence and grade of vesicoureteral reflux

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years
* Undergoing endoscopic urological surgery
* With or without a prior VCUG performed for urinary tract infection or other clinical indications
* Availability of VCUG results for participants who previously underwent VCUG
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* History of previous ureteral reimplantation or anti-reflux surgery
* Known neurogenic bladder or severe lower urinary tract dysfunction
* Active urinary tract infection at the time of endoscopic procedure
* Inability to undergo fluoroscopic imaging (e.g., contrast allergy)
* Incomplete clinical or imaging data

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Detection of vesicoureteral reflux (VUR) by PIC cystography compared with VCUG | During endoscopic surgery (single intraoperative assessment)
  Detection of vesicoureteral reflux (VUR) by PIC cystography compared with VCUG, assessed as the presence or absence of reflux and categorized as low-grade (Grade 1-3) or high-grade (Grade 4-5) on a renal unit basis.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Urology Department, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided